CLINICAL TRIAL: NCT01344590
Title: Ethanol Lock for Prevention of Central Line-Associated Blood Stream Infections
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Virginia (Other)
Responsible Party: Ronald Truner, MD, University of Virginia
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: 15397
Record Dates: First submitted 2011-04-27; First posted 2011-04-29 (Estimated); Last update posted 2011-04-29 (Estimated); Status verified 2011-04

CONDITIONS: Central Lines in ICU Patients
Keywords: central line associated blood stream infections
MeSH Terms: interventions — Saline Solution; Ethanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- saline lock maintenance (Active Comparator): Standard saline lock maintenance
  Interventions: Other: Normal Saline
- ethanol maintenance (Experimental): Instillation of 70% pharmaceutical grade ethanol solution into the central line in a volume calculated to fill the catheter lumen and hub.
  Interventions: Other: Ethanol 70% pharmaceutical grade

INTERVENTIONS:
Other: Normal Saline — Standard saline procedure will be utilized.
  Arms: saline lock maintenance
Other: Ethanol 70% pharmaceutical grade — 70% pharmaceutical grade ethanol will be instilled in the line in a volume calculated to fill the lumen and the hub.
  Arms: ethanol maintenance

SUMMARY:
Vascular access via central venous lines (CVL) is essential to the care of many patients in the intensive care setting. While the value of these lines for the management of critically ill patients is generally accepted, the potential for line-associated blood stream infection is a known complication of the use of this intervention.

Ethanol is an effective antimicrobial agent with activity against a broad spectrum of human pathogens.

The purpose of this study is to evaluate the effectiveness of daily treatment of the catheter lumen with ethanol to prevent central line associated blood stream infections (CLABSI). The hypothesis is that this treatment will reduce the incidence of CLABSI compared to maintenance of the lines with normal saline alone.

DETAILED DESCRIPTION:
Blood stream infections are an important complication of the use of central venous lines (CVLs) and result in increased morbidity, mortality, and cost. Blood stream infections related to CVLs may be the result of migration of skin organisms along the catheter tract or introduction of organisms into the lumen of the catheter. The extraluminal route of infection appears to be most common early after catheter insertion while the frequency of infection acquired by the intraluminal route appears to increase the longer the catheter is in place. Meticulous attention to best practices for insertion and the subsequent care of the insertion site reduces infection by the extraluminal route. Adherence to good technique for entering the line may similarly reduce infection by the intraluminal route.

Ethanol is an effective antimicrobial agent with activity against a broad spectrum of human pathogens; including the bacteria and fungi which most commonly infect CVLs. The mechanism of the antimicrobial activity of ethanol is attributed to the ability to denature proteins and induced resistance to the effect of ethanol has not been reported. These features suggest that ethanol-lock is a promising approach to the prevention of acquisition of central line associated blood stream infections by the intraluminal route.

ELIGIBILITY:
Although this study is done in the patient-care setting, patients are not the subject of the study. The outcome of interest involves the development of CLABSI in patients but the intervention is directed at the patient's central lines rather than the patient. There are no inclusion or exclusion criteria; the determination of the line care regimen will be determined by the bed assignment rather than any characteristics of the patient occupying the bed.

All central line will be included in this study. Use of ethanol will be suspended whenever the usage of the line precludes instillation of ethanol with a dwell time of al least one hour.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2011-02; Primary Completion 2012-05 (Estimated); Study Completion 2012-05 (Estimated)

PRIMARY OUTCOMES:
Number of beds using ethanol treatment | 12 months
  The primary endpoint of the study will be the effectiveness of ethanol for prevention of CLABSI compared to routine care. This will be assessed at the end of the study (12 months)by comparing the number of beds being maintained by each regimine to determine if the distribution of line maintenance regimines is non-random in favor of either ethanol lock or saline maintenance.

CONTACTS AND LOCATIONS:
Overall Officials: Ron Turner, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States